CLINICAL TRIAL: NCT04758637
Title: Application of Economics & Social Psychology to Improve Opioid Prescribing Safety Trial 2 (AESOPS-2): Availability of Opioid Harm
Brief Title: AESOPS Trial 2 (AESOPS-2): Availability of Opioid Harm
Acronym: AESOPS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Northwestern University (Other); AltaMed Health Services Corporation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UP-20-01330; R33AG057395 (NIH)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Opioid Abuse
Keywords: opioid use disorder; randomized control trial; behavioral economics; nudges
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Physicians in the control group will receive no notification of their patient's fatal or nonfatal overdose.
- Overdose Notification Group (Experimental): The overdose notifications will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses.
  Interventions: Behavioral: Overdose Notification

INTERVENTIONS:
Behavioral: Overdose Notification — We will identify overdoses from state vital records and insurance claims data linked to emergency departments. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a non-fatal or fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the deceased or surviving patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
  Arms: Overdose Notification Group

SUMMARY:
The opioid epidemic is the largest man-made public health crisis the United States has faced. The objective of Trial 2 of the Application of Economics & Social psychology to improve Opioid Prescribing Safety (AESOPS-2) study, is to discourage unnecessary opioid prescribing by increasing the salience of negative patient outcomes associated with opioid use.

DETAILED DESCRIPTION:
In AESOPS-2, a multi-site study, random assignment determines if prescribers to persons who suffer an opioid overdose (fatal or nonfatal) learn of this event (intervention) or practice usual-care (control). The AESOPS-2 trial will take place in 3 diverse health systems in the U.S. - Northwestern Medicine, AltaMed Health Services, and The Children's Clinic. At Northwestern Medicine, clinicians in the intervention group receive a letter notifying them of their patient's fatal or nonfatal ED overdose. At AltaMed Health Services, and The Children's Clinic, clinicians in the intervention group receive a letter notifying them of their patient's nonfatal ED overdose. The primary outcome is the change in clinician weekly milligram morphine equivalent (MME) dose prescribed in 6-month periods before and after receiving the letter. The secondary outcome is the change in the proportion of patients prescribed at least 50 daily MME. Group differences in these outcomes will be compared using an intent-to-treat difference-in-differences framework with a mixed-effects regression model to estimate clinician MME weekly dose. The AESOPS-2 trial will provide new knowledge about whether increasing prescribers' awareness of patients' opioid-related overdoses leads to a reduction in opioid prescribing. Additionally, this trial may better inform how to reduce opioid use disorder and opioid overdoses by lowering unnecessary population exposure to these drugs.

ELIGIBILITY:
Inclusion Criteria:

* 1) The clinician prescribed a qualifying scheduled drug to a patient in the 12 months prior to their non-fatal or fatal overdose 2) the patient is 18 years old or older at the time of the overdose, 3) the provider practices within a health system enrolled in the study, and 4) the overdose occurs during the 12-month observation period. Qualifying prescriptions include those for one of the following scheduled drugs: opioids, benzodiazepines, muscle relaxants or sedative-hypnotics.

Exclusion Criteria:

* Prescriptions to patients in hospice or with active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kelley MA, Persell SD, Linder JA, Friedberg MW, Meeker D, Fox CR, Goldstein NJ, Knight TK, Zein D, Sullivan MD, Doctor JN. The protocol of the Application of Economics & Social psychology to improve Opioid Prescribing Safety trial 2 (AESOPS-2): Availability of opioid harm. Contemp Clin Trials. 2022 Jan;112:106650. doi: 10.1016/j.cct.2021.106650. Epub 2021 Dec 8. PMID 34896295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prescriber did or did not receive the letter based on the randomization assignment (intervention or control) of the overdose victim. Clinician prescribing data was collected during the study timeframe.
Pre-assignment Details: Patients who experienced an opioid overdose were randomized to either the letter intervention (fatal or non fatal overdose) or control; however, patients were not considered enrolled in the study. We analyze how the prescribing behavior of clinicians who had prescribed opioids to these patients changed pre-to-post intervention.
Groups:
- Nonfatal Control Group: Physicians in the nonfatal control group will receive no notification of their patient's nonfatal overdose.
- Non Fatal Overdose Notification Group: Non Fatal Overdose Notification: We will identify overdoses from insurance claims data linked to emergency departments. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a non-fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
- Fatal Control Group: Physicians in the fatal control group will receive no notification of their patient's fatal overdose.
- Fatal Overdose Notification Group: Fatal Overdose Notification: We will identify overdoses from state vital records. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the deceased patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
Period: Overall Study
Arm/Group | Nonfatal Control Group | Non Fatal Overdose Notification Group | Fatal Control Group | Fatal Overdose Notification Group
Started | 19 | 20 | 11 | 11
Patient Overdose Victims | 16 | 14 | 10 | 10
Completed | 19 | 19 | 11 | 11
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non Fatal Control Group: Physicians in the non fatal control group will receive no notification of their patient's nonfatal overdose.
- Non Fatal Overdose Notification Group: Non Fatal Overdose Notification: We will identify overdoses from insurance claims data linked to emergency departments. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a non-fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the deceased or surviving patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
- Fatal Overdose Notification Group: Fatal Overdose Notification: We will identify overdoses from state vital records. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the deceased or surviving patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
- Total: Total of all reporting groups
Arm/Group | Non Fatal Control Group | Non Fatal Overdose Notification Group | Fatal Control Group | Fatal Overdose Notification Group | Total
Number analyzed (Participants) | 19 | 20 | 11 | 11 | 61
Age, Customized [Count of Participants; unit: Participants] — Age data not collected. Population: Age data not collected.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 11 | 5 | 2 | 27
  Male | 8 | 9 | 6 | 9 | 32
  Missing | 2 | 0 | 0 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 11 | 11 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Average Number of 5 MME Pill Counts
Description: The primary outcome is the change in daily average number of 5 morphine milligram equivalent (MME) pill counts ordered by clinicians during the last week of baseline (week 26) and the last week of the intervention period (week 53) letter intervention.
Time Frame: 13 months (6 months pre-intervention, 30-day washout period, 6 months post-intervention)
Population: Participating clinicians from Northwestern Medicine and AltaMed who prescribed an opioid during the study period
Measure: Mean (95% Confidence Interval); unit: Difference in estimated mean pill counts
Arm/Group | Non Fatal Control Group | Non Fatal Overdose Notification Group | Fatal Control Group | Fatal Overdose Notification Group
Number analyzed (Participants) | 19 | 19 | 11 | 11
Difference in estimated mean pill counts | -3.73 [-6.00 to -0.79] | 3.89 [1.61 to 7.58] | 9.8 [3.86 to 18.9] | -4.85 [-6.24 to -3.11]
Statistical Analysis 1: Comparison: Non Fatal Control Group vs Non Fatal Overdose Notification Group; Null hypothesis is the difference in difference in estimated mean pill counts from the last week of baseline (week 26) to the last week of the intervention period (week 53) between control and non-fatal is 0; Test type: Superiority; p = 0, Zero-inflated Poisson mixed regression — The calculated p-value is 7.62E-10; Model estimates were used to derive estimated difference in difference value. Confidence intervals were bootstrapped using 1000 repetitions; Mean Difference (Final Values) = 7.62, 95% CI 2-sided [2.4 to 13.59]
Statistical Analysis 2: Comparison: Fatal Control Group vs Fatal Overdose Notification Group; Null hypothesis is the difference in difference in estimated means from the study start (week 0) to the study end (week 23) between control and fatal is 0; Test type: Superiority; p = 0, Zero-inflated Poisson mixed regression — The calculated p-value is 2E-16; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.65, 95% CI 2-sided [-25.14 to -6.97]

2. Secondary Outcome: Change in Clinician-level, Pre-to-post Mean Proportion of High Dose (=> 50 MME) Patient Visits
Description: The change in the clinician-level, pre-to-post mean proportion of high dose (=> 50 MME) patient visits by study arm. The numerator is whether a patient visit was => 50 MME, and the denominator is the number of opioids. We quantified this measure using logistic regression. Higher dose prescriptions are not recommended and are associated with the potential for greater patient harm.
Time Frame: 13 months (6 months pre-intervention, 30-day washout period, 6 months post-intervention)
Measure: Mean (95% Confidence Interval); unit: proportion of high dose patient visits
Arm/Group | Non Fatal Control Group | Non Fatal Overdose Notification Group | Fatal Control Group | Fatal Overdose Notification Group
Number analyzed (Participants) | 19 | 19 | 11 | 11
proportion of high dose patient visits | 0.004 [-0.012 to 0.045] | 0.014 [-0.001 to 0.098] | 0.01 [-0.06 to 0.15] | -0.09 [-0.12 to 0.07]
Statistical Analysis 1: Comparison: Non Fatal Control Group vs Non Fatal Overdose Notification Group; Test type: Superiority; p = 0.219, Regression, Logistic; Slope = 0.72, 95% CI 2-sided [-0.43 to 1.86]
Statistical Analysis 2: Comparison: Fatal Control Group vs Fatal Overdose Notification Group; Test type: Superiority; p = 0.229, Regression, Logistic; Slope = -0.72, 95% CI 2-sided [-1.9 to 0.46]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event collection is based on the patients of randomized clinicians, not the clinicians themselves. Deaths and adverse events were not collected for clinicians.
Groups:
- Non Fatal Control Group: Physicians in the non fatal control group will receive no notification of their patient's non fatal overdose.
- Non Fatal Overdose Notification Group: The overdose notifications will alert prescribers to the patient's opioid-related non fatal overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses.
  Overdose Notification: We will identify overdoses from insurance claims data linked to emergency departments. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a non-fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the surviving patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
- Fatal Overdose Notification Group: The fatal overdose notifications will alert prescribers to the patient's fatal opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses.
  Overdose Notification: We will identify overdose deaths from state vital records. We will use electronic health record data to identify prescriptions of scheduled drug to patients who experienced a fatal overdose within the health system. If randomized to the overdose notification group, physicians who prescribed the controlled substances to the deceased patient in the year prior to their overdose will be informed of the overdose via letter. The letters will alert prescribers to the patient's opioid-related overdose, recommend the use of the state-level PDMP, and list evidence-based interventions to lower opioid-related overdoses. The letters will increase the salience and availability of opioid-related harms, which may cause clinicians to be more wary of a future overdose when prescribing opioids, benzodiazepines, muscle relaxants, or sedative-hypnotics.
Arm/Group | Non Fatal Control Group | Non Fatal Overdose Notification Group | Fatal Control Group | Fatal Overdose Notification Group
All-Cause Mortality (participants affected / at risk) | 0/861 | 0/973 | 0/524 | 0/801
Serious Adverse Events (participants affected / at risk) | 1/861 | 1/973 | 1/524 | 0/801
Other Adverse Events (participants affected / at risk) | 0/861 | 0/973 | 0/524 | 0/801
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Fatal Control Group (N=861) | Non Fatal Overdose Notification Group (N=973) | Fatal Control Group (N=524) | Fatal Overdose Notification Group (N=801)
Emergency Department or Hospitalization for Opioid Withdrawal (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 — Emergency Department or Hospitalization for Opioid Withdrawal for any patients of randomized clinicians with an opioid prescription in the 6 month post-intervention period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT04758637/Prot_SAP_000.pdf